CLINICAL TRIAL: NCT01807676
Title: Prospective, Randomized Clinical Trial Evaluating the ETView Double-Lumen Tube
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0520
Record Dates: First submitted 2013-03-07; First posted 2013-03-08 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Patients Undergoing Elective Thoracic Surgery Requiring Obligatory Single-lung Ventilation During Surgery

ARMS (2):
- ET View Double Lumen Tube (Active Comparator): Patients assigned to the thisgroup will be intubated using the VivaSight-DL.
  Interventions: Device: ET View Double Lumen Tube
- conventional Double Lumen Tube (Active Comparator): Patients assigned to the first group will be intubated using conventional DLT (Bronchocath, left sided; Rüsch, Kernen, Germany).
  Interventions: Device: conventional Double Lumen Tube

INTERVENTIONS:
Device: ET View Double Lumen Tube
  Other Names: VivaSight-DL (ETView Ltd, M.P. Misgav 20174, Israel)
  Arms: ET View Double Lumen Tube
Device: conventional Double Lumen Tube
  Other Names: conventional DLT (Bronchocath, left sided; Rüsch, Kernen, Germany)
  Arms: conventional Double Lumen Tube

SUMMARY:
No prospective randomized clinical trial assessed the performance of this new device in a clinical setting. Consequently the aim of this study is to determine clinical performance of this new device compared with conventional DLT.

* Trial with medical device

DETAILED DESCRIPTION:
In several clinical situations and surgical procedures single-lung ventilation (SLV) is essential. Especially during thoracic surgery SLV and collapse of the operated lung, while ventilating the other side of the lung is the most frequented indication. In these cases the double lumen tube (DLT) is the most widely used device.

The DLT consists of a proximal tracheal and a distal bronchial end, reaching into the left or the right side of the lung- dependent of the model of the tube. Endotracheal intubation with DLT, which are much larger and stiffer than conventional single-lumen tubes, are much more difficult to place and are especially likely to provoke airway injuries. Furthermore, placement of a DLT requires obligatory fiberoptic bronchoscopy and a certain level of experience. Tube misplacement after patients removal from dorsal (intubation-) to lateral position as well as during surgical procedure is relatively frequent. Tube displacement from its proper position above the carina, respectively in the main bronchus, may result in life-threating complications and airway lacerations.

The anesthetist may detect tube misplacement from indirect clinical signs including increased airway pressure, oxygen desaturation, or difficulty performing SLV. In this clinical situations, verification of tube position using fibreoptic bronchoscopy is indicated. Fibreoptic bronchoscopy requires rigorous training and practice to maintain a high level of skill as well as expensive infrastructure.

The VivaSight-DL (ETView Ltd, M.P. Misgav 20174, Israel) is a new DLT promising to exceed clinical performance of the conventional DLT. The VivaSight-DL is basically a left-sided DLT with an embedded video imaging device and light source at its tip and integrated cable with connector. However, after correct tube placement, the video imaging device is focused on the main carina, indicating the correct position of the bronchial cuff in the left main bronchus.

ELIGIBILITY:
Inclusion criteria:

* Elective thoracic surgery with anticipated use of a DLT
* Anticipated extubation in the operating room;
* American Society of Anesthesiologist Physical Status 1-3;
* Age 18- 90.
* Written consent (signature from patient)

Exclusion criteria:

* Tracheal pathology, including tracheostomy;
* Any form of infection (including upper-respiratory tract infection or pneumonia) or suspected tuberculosis;
* BMI higher exceeding 40 kg/m2;
* Known or suspected difficult airway.
* Pregnancy
* Breast feeding
* The subject must not be involved in any other clinical trial during the course of this trial, nor within a period of 30 days prior to its beginning or 30 days after its completion

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-03; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
time to intubation | 300 seconds
  Time for intubation, defined as "time from insertion of the laryngoscope until statement of the intubating anesthesiologist, that DLT was correctly placed". Time for intubation will be measured by an independent researcher using a stop watch.

SECONDARY OUTCOMES:
Rate of misplacement | 3 hours
  Rate of misplacement, occurring after patients removal from dorsal to lateral position
Rate of misplacement | 3 hours
  Rate of misplacement, occurring during surgery, potentially caused by vibrations and movements by surgeons
Rate of blind insertion | 300 seconds
  Rate of blind insertion, defined as successful placement of airway device in correct position in trachea/ main stream bronchus without help of fibreoptic bronchoscopy8
rate of fibreoptic bronchoscopy | 3 hours
  Necessity of tube re-placement by fibreoptic bronchoscopy
Quality of lung collapse | 3 hours
Airway injuries | 3 hours
Postoperative coughing | 24 hours
Postoperative hoarseness | 24 hours
Postoperative sore throat | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice Beck Schimmer, Prof MD, Principal Investigator — University Hospital Zurich, Division of Anaesthesiology
Locations (1):
- University Hospital Zurich, Division of Anaesthesiology, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Schuepbach R, Grande B, Camen G, Schmidt AR, Fischer H, Sessler DI, Seifert B, Spahn DR, Ruetzler K. Intubation with VivaSight or conventional left-sided double-lumen tubes: a randomized trial. Can J Anaesth. 2015 Jul;62(7):762-9. doi: 10.1007/s12630-015-0329-8. Epub 2015 Feb 6. PMID 25663254